CLINICAL TRIAL: NCT02609490
Title: A Multi-center, Randomized, Double-blind, Double-dummy, With Olmesartan Medoxomil as Positive Control Parallel Clinical Study to Evaluate the the Safety and Efficacy of Azilsartan in Chinese Patients With Primary Mild and Moderate Hypertension
Brief Title: Azilsartan in Chinese Patients With Mild and Moderate Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Zhaoke-201505-Azilsartan
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — azilsartan; Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment-Azilsartan (Experimental): Azilsartan tabelts
  Interventions: Drug: Azilsartan tablets; Drug: olmesartan medoxomil placebo tablets
- Positive Control-olmesartan medoxomil (Active Comparator): olmesartan medoxomil tablets
  Interventions: Drug: Azilsartan placebo tablets; Drug: Olmesartan medoxomil tablets

INTERVENTIONS:
Drug: Azilsartan tablets — 20mg/tablet
  Arms: Treatment-Azilsartan
Drug: Azilsartan placebo tablets — placebo tablet
  Arms: Positive Control-olmesartan medoxomil
Drug: Olmesartan medoxomil tablets — 20mg/tablet
  Arms: Positive Control-olmesartan medoxomil
Drug: olmesartan medoxomil placebo tablets — placebo tablet
  Arms: Treatment-Azilsartan

SUMMARY:
A phase 3 clinical study to evaluate the safety and efficacy of Azilsartan in Chinese hypertension patients

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years of age (including 18 and 70 years of age), male or female;
2. diagnosed with mild to moderate essential hypertension;
3. clinic diastolic and systolic blood pressure need to meet the following two conditions: 3 times mean sitting diastolic blood pressure measurements at 95mmHg-110mmHg (not including 110mmHg); 3 times sitting systolic blood pressure measured and mean value between150mmHg-180mmHg (not including 180mmHg);
4. understand clearly that voluntary to participate in the study, sign informed consent.

Exclusion Criteria:

1. severe essential hypertension (sitting systolic ≥180mmHg and / or sitting diastolic pressure ≥110mmHg), malignant hypertension, hypertensive emergency, hypertensive crisis and high blood pressure encephalopathy.
2. secondary hypertension.
3. The following hypertension and diseases: acute myocardial infarction within 6 months, the cerebral artery accident, transient ischemic attack; or dissecting aortic aneurysm, angina, II-IVClass (NYHA classification) history of heart failure Ⅱ degree atrioventricular block, sick sinus integrated disease, bradycardia (heart rate <50 beats / min) or other antiarrhythmic drugs needed.
4. significant laboratory abnormalities include: serum potassium> 5.5mmol / L; blood ALT or AST> 2.5ULN; serum creatinine> 1.5ULN.
5. unilateral or bilateral renal artery stenosis.
6. Type 1 diabetes and poor glycemic control of type 2 diabetes (HbA1c values ≥ 8%).
7. gastrointestinal lesions or gastrointestinal surgery may affect drug absorption or excretion, such as stomach-bowel resection, nearly one year activity of gastrointestinal inflammation, ulcers or gastrointestinal bleeding.
8. azilsartan sheet or olmesartan medoxomil tablets and related drugs (ARB, ACEI And renin inhibitors) allergies.
9. pregnant, lactating female patients, or during the test does not guarantee the effective collision pregnant person.
10. Obesity, body mass index (BMI)> 30kg / m2.
11. Import of use in addition to import other types of medication trials of antihypertensive drugs, Anti-angina drugs, lithium agents, corticosteroids, licorice, estrogen, digitalis Drugs and drugs were potassium.
12. Variance of diastolic blood pressure ≥8mmHg.
13. drug or alcohol abuse within 6 months Are drinking more than two units of alcohol (1 unit = 360mL or 45mL alcohol content of 40%).

14 patients with malignant tumors. 15. hemodialysis patients or strictly limit salt therapy. 16. Participated in other clinical trials within 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Decrease of sitting diastolic blood pressure at week 16 | 16 weeks

SECONDARY OUTCOMES:
Decrease of sitting diastolic blood pressure at week 8 | 8 weeks
Decrease of sitting systolic blood pressure at week 8 | 8 weeks
Decrease of sitting diastolic blood pressure at week 2 | 2 weeks
Decrease of sitting diastolic blood pressure at week 4 | 4 weeks
Decrease of sitting diastolic blood pressure at week 12 | 12weeks
Decrease of sitting systolic blood pressure at week 2 | 2 weeks
Decrease of sitting systolic blood pressure at week 4 | 4 weeks
Decrease of sitting systolic blood pressure at week 12 | 12 weeks
decrease of 24-hour ambulatory blood pressure monitoring at week 16 | 16 week
  do a 24-hour ambulatory blood pressure monitoring at baseline and at week 16, compare the decrease.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First hospiatl, Beijing, China